CLINICAL TRIAL: NCT05278598
Title: Comparative Assessment of 3 Ultrasound Guided Plane Blocks for Perioperative Analgesia in Patients Undergoing Radical Cystectomy: A Randomized Clinical Trial
Brief Title: 3 Ultrasound Guided Plane Blocks for Perioperative Analgesia in Patients Undergoing Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3USGPBPORC
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cancer, Bladder; Surgery; Anesthesia; Analgesia; Block
Keywords: Erector spinae plane block; Quadratus lumborum plane block; Paravertebral block; Ultrasound-guided; Radical cystectomy; Analgesia; Anesthesia
MeSH Terms: conditions — Urinary Bladder Neoplasms; Agnosia; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESPB group (Active Comparator): Erector Spinae Plane Block
  Interventions: Procedure: Erector Spinae Plane Block
- TPVPB group (Active Comparator): Thoracic Paravertebral Plane Block
  Interventions: Procedure: Thoracic Paravertebral Plane Block
- QLPB group (Active Comparator): Quadratus Lumborum Plane Block
  Interventions: Procedure: Quadratus Lumborum Plane Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — After skin sterilization, ESP block will be performed at the level of T9. A curvilinear high-frequency ultrasound transducer will be placed sagittal 3 cm lateral to T9 spinous process where a hyperechoic shadow of the transverse process (TP) and erector spinae will be defined. A 22-gauge spinal needle will be inserted in cranial to caudal direction toward TP in plane to the ultrasound transducer until the needle touches the TP crossing the whole muscles. The location of the needle tip will be confirmed by visible normal saline solution separating erector spinae muscle off the bony shadow of the TP on ultrasound imaging. After confirming the needle site, 30 mL of 0.25% bupivacaine will be injected. Sonographic confirmation of the local anesthetic spread will be seen as an anechoic shadow in the paravertebral spaces from T7 to T12.
  This procedure will be done on both sides.
  Arms: ESPB group
Procedure: Thoracic Paravertebral Plane Block — After skin sterilization, curvilinear high-frequency ultrasound transducer will be used to visualize the T10 paravertebral space in the paramedian sagittal plane. An injection into the paravertebral space will spread to multiple adjacent dermatomes, so exact identification of a specific level will be not necessary. A 22-gauge spinal needle will be inserted in-plane relative to the ultrasound probe and slowly be directed from lateral to medial until its tip was located at the apex of the paravertebral space and the endpoint for successful block will be anterior displacement of the pleura by injected local anesthetic where a single injection of 30 ml of 0.25% bupivacaine will be injected.
  This procedure will be done on both sides.
  Arms: TPVPB group
Procedure: Quadratus Lumborum Plane Block — After skin sterilization, curvilinear high-frequency ultrasound transducer will be positioned horizontally in the anterior axillary line halfway between the subcostal margin and iliac crest, to locate the triple abdominal muscle layers, then the probe will be relocated subsequently to the posterior axillary line until the quadratus lumborum muscle could be visualized with its attachment to the lateral edge of the transverse process of the L4 vertebral body. With the psoas major muscle anteriorly, the erector spinae muscle posteriorly and the quadratus lumborum muscle adherent to the apex of the transverse process, this is a well-recognizable pattern of a shamrock with three leaves. A 22-gauge spinal needle will be inserted in-plane relative to the ultrasound probe passing in posterior to anterior direction through the quadratus lumborum to reach the border between it and psoas major, where 30 ml of 0.25% bupivacaine will be injected.
  This procedure will be done on both sides.
  Arms: QLPB group

SUMMARY:
Radical cystectomy is the gold standard treatment for muscle invasive bladder cancer as well as some T1 and non-invasive disease. It is a major operation with significant perioperative morbidity and complications. Pain is one of the most important complications to be managed.

Regional blocks as a part of multi-modal analgesia are considered main strategies of Enhanced Recovery after Surgery (ERAS) decreasing post-operative complications including post-operative pain and post-operative hospital stay. They also have an upper hand over systemic intravenous opioids decreasing the risk for post-operative delirium specially in old age patients. Thoracic paravertebral plane block (TPVPB), intra muscular quadratus lumborum plane block (QLPB) and erector spinae plane block (ESPB) are among these regional anesthesia techniques for pain management.

Erector spinae plane block is an emerging block, with low risk and more feasibility, but efficacy hasn't been compared to quadratus lumborum and paravertebral plane blocks altogether in radical cystectomy surgeries.

All these blocks are effective in reducing postoperative pain and the need of analgesia in radical cystectomy surgery; this is a comparative study between the three blocks in this population.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class II - III.
* Adult patients scheduled for radical cystectomy.

Exclusion Criteria:

* Patient refusal.
* Uncooperative patients.
* Patients with known allergies to local anesthetics.
* Bleeding disorders or coagulopathy.
* Anatomical abnormality or infection at injection site.
* Patients receiving opioids for chronic analgesic therapy.
* Spinal anesthesia or any other regional anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Morphine consumption. | 24 hours
  Total dose of Morphine (measured in mg) given intra-venously to the patient post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa M Zalat, MSc, Principal Investigator — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Nazmy S Michael, MD, Study Director — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt